CLINICAL TRIAL: NCT03338322
Title: Postoperative Pain After Using Reciprocating Motion With Reciproc Files Versus Adaptive Motion With Twisted File Adaptive In Instrumentation Of Necrotic Mandibular Molars: A Randomized Clinical Trial
Brief Title: Postoperative Pain After Using Reciprocating Motion With Reciproc Files Versus Adaptive Motion With Twisted File Adaptive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Yaser Abu Bakr, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: twisted file adaptive 1987
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; reciproc; twisted file adaptive
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Twisted file adaptive (Experimental): Files that are used in root canal preparation in adaptive motion
  Interventions: Device: Twisted file adaptive
- Reciproc (Active Comparator): Reciproc files are used in root canal preparation with reciprocation motion
  Interventions: Device: Reciproc

INTERVENTIONS:
Device: Twisted file adaptive — Endodontic files that are used in preparation of root canals with adaptive motion
  Arms: Twisted file adaptive
Device: Reciproc — Endodontic files that are used in root canal preparation with reciprocation motion
  Arms: Reciproc

SUMMARY:
assess the effect of using reciprocating motion with reciproc files versus adaptive motion using twisted file adaptive on postoperative pain after instrumentation of necrotic mandibular molars.

DETAILED DESCRIPTION:
In root canal treatment of mandibular molar teeth in patients having necrotic pulp with symptomatic or asymptomatic apical periodontitis, Is there difference in postoperative pain after instrumentation between two different kinematics; adaptive motion using Twisted File Adaptive and reciprocation motion using Reciproc

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are medically free from any systemic disease that may contraindicate our interventions.
2. Patient's age between 18-60 years old.
3. Mandibular molars having necrotic pulps with symptomatic or asymptomatic apical periodontitis because this group of patients may have more postoperative pain than vital teeth22.
4. Positive patient's acceptance for participation in the study.

Exclusion Criteria:

1. Patients who had used any type of analgesic medication during the preceding 12 hours before the treatment to give true response of pain after instrumentation.
2. Teeth with vital pulps or Symptomatic irreversible pulpitis.
3. Pregnant patients or lactating because of radiographic hazards and use of analgesics27.
4. Any known sensitivity or adverse reactions to ibuprofen.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Post instrumentation pain | up to 7 days
  post instrumentation pain will be recorded by the patient using numerical rating scale (0-10) will be used to record pain intensity

SECONDARY OUTCOMES:
analgesic intake | up to 7 days
  number of analgesic intake will be recorded by the patient
Colony forming units | 6 hours
  calculation of colony forming units before and after instrumentation

IPD SHARING:
Plan to Share IPD: Undecided
participant data will be recorded and shared